CLINICAL TRIAL: NCT02820740
Title: Feasibility Study on Laser Interstitial Thermal Therapy Ablation for the Treatment of Medical Refractory Epilepsy (FLARE)
Brief Title: Feasibility Study on LITT for Medical Refractory Epilepsy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated (failure to enroll)
Sponsor: Monteris Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLARE
Record Dates: First submitted 2016-06-08; First posted 2016-07-01 (Estimated); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-05

CONDITIONS: Epilepsy
Keywords: Epilepsy; Medial Temporal Lobe Epilepsy; Seizure; NeuroBlate; LITT; Quality of Life
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- NeuroBlate LITT Treatment (Other): This is a single arm study. All eligible study subjects will undergo LITT with the NeuroBlate System.
  Interventions: Device: NeuroBlate System

INTERVENTIONS:
Device: NeuroBlate System — Laser Interstitial Thermal Therapy

SUMMARY:
Multicenter, open-label, prospective designed study to characterize the performance of brain laser interstitial thermal therapy (LITT) ablation using the Monteris NeuroBlate System for the treatment of drug-refractory medial temporal lobe epilepsy in subjects who are candidates for LITT surgery.

DETAILED DESCRIPTION:
Monteris is sponsoring this multicenter, open-label, prospective feasibility study to characterize the performance of laser interstitial thermal therapy (LITT) using the Monteris NeuroBlate System for the treatment of drug-refractory medial temporal lobe epilepsy in subjects who are candidates for LITT surgery.

The NeuroBlate System uses precise, high-intensity laser light to initiate necrosis of abnormal brain tissue through thermal ablation while limiting injury to healthy tissue. Unlike traditional brain surgery, LITT does not require a large opening in the skull.

Subjects who meet the study eligibility criteria and sign the informed consent form will undergo the LITT procedure. Subjects, or their caregivers, are required to keep a seizure diary throughout the study, beginning after surgery. The study will monitor and record subjects' seizure frequency, antiepileptic medications, and physical and emotional health.

Subjects treated with NeuroBlate will have 2 years of follow-up. Throughout study participation, the study investigator will continuously monitor and document both effectiveness and safety data at study appointments.

ELIGIBILITY:
Relevant Inclusion Criteria are listed below

* Diagnosis of unilateral medial temporal lobe epilepsy (MTLE) confirmed clinically and with either (1) ictal scalp recording and MRI evidence of mesial temporal sclerosis or (2) intracranial ictal onset consistent with hippocampal origin
* Averages 1 or more complex partial seizures or secondary generalized seizures compatible with MTLE per month
* On stable antiepileptic medications
* Meets the criteria for a medial temporal lobe resection and is a candidate for LITT
* 18 years or older at the time of consent

Relevant Exclusion Criteria are listed below

* Previous diagnosis of psychogenic/non-epileptic seizures
* Previous diagnosis of primary generalized seizures
* IQ less than 70
* Subject has a MRI-incompatible implanted electronic device or any metallic prosthesis or implant for which brain MRI is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Spencer, MD, Principal Investigator — Yale University
Locations (5):
- United States (5):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mount Sinai West, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- NeuroBlate LITT Treatment: All eligible study subjects who underwent LITT with the NeuroBlate System.
Period: Overall Study
Arm/Group | NeuroBlate LITT Treatment
Started | 4
Completed | 2
Not Completed | 2
Not completed — Did not have procedure | 2

BASELINE CHARACTERISTICS:
Arm/Group | NeuroBlate LITT Treatment
Number analyzed (Participants) | 2
Age, Customized [Median (Full Range); unit: years]
  Age range | 55 [53 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Characterize adverse events experienced in medial temporal lobe epilepsy subjects undergoing LITT using the NeuroBlate System. Adverse events will be collected based on subject reports and subject examination/testing.
Time Frame: 2 Years
Population: The per-protocol analysis was not completed because the study was terminated early and the data collected was insufficient for the analysis despite two subjects completing the study at 24 months.
Measure: Count of Participants; unit: Participants
Arm/Group | NeuroBlate LITT Treatment
Number analyzed (Participants) | 2
Participants | 2

2. Primary Outcome: Changes in Neuropsychological Functioning
Description: Characterize changes to neuropsychological functioning experienced in medial temporal lobe epilepsy subjects undergoing LITT using the NeuroBlate System. Descriptive statistics (via neuropsychological assessment tools) will be reported for the measured score at baseline and each follow-up visit.
Time Frame: 1 Year
Population: The per-protocol analysis was not completed because the study was terminated early and the data collected was insufficient for the analysis.
Measure: Mean (Full Range); unit: Time in seconds
Arm/Group | NeuroBlate LITT Treatment
Number analyzed (Participants) | 2
Time in seconds
  Baseline Trails Making Trial A | 29.5 [24 to 35]
  Baseline Trails Making Trial B | 66 [47 to 85]
  1 Year Trails Making A | 32.5 [26 to 39]
  1 Year Trails Making B | 59.5 [43 to 76]

3. Secondary Outcome: Changes in Seizure Frequency
Description: Characterize changes in seizure frequency experienced in medial temporal lobe epilepsy subjects undergoing LITT using the NeuroBlate System by utilizing patient diary to evaluate seizure occurrences.
Time Frame: 2 Years
Population: as for outcome 2
Measure: Median (Full Range); unit: Number of seizures/month
Arm/Group | NeuroBlate LITT Treatment
Number analyzed (Participants) | 2
Number of seizures/month
  Seizures at baseline | 22 [8 to 34]
  Seizures at 24 Months | 3 [0 to 6]

4. Secondary Outcome: Surgical Outcome Classification
Description: Characterize the Engel and ILAE surgical outcome classification in medial temporal lobe epilepsy subjects undergoing LITT using the NeuroBlate System. Classifications will be determined by the Investigator.
  Engel Scale Class I: Free of disabling seizures Class II: Rare disabling seizures Class III: Worthwhile improvement Class IV: No worthwhile improvement
  ILAE Outcome Scale Class 1: Completely seizure free; no auras Class 2: Only auras; no other seizures Class 3: 1 to 3 seizure days per year; ± auras Class 4: 4 seizure days per year to 50% reduction of baseline seizure days; ± auras Class 5: Less than 50% reduction of baseline seizure days; ± auras Class 6: More than 100% increase of baseline seizure days; ± auras
Time Frame: 2 Years
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | NeuroBlate LITT Treatment
Number analyzed (Participants) | 2
participants
  Engel Class III at 2 years | 1
  Engel Class I at 2 years | 1
  ILAE Class 4 at 2 years | 1
  ILAE Class 1 at 2 years | 1

5. Secondary Outcome: Changes in Quality of Life
Description: Characterize the changes in quality of life in subjects with medical temporal lobe epilepsy undergoing LITT using the NeuroBlate System. Quality of life will be measured using the QOLIE-31 (Quality of Life in Epilepsy) questionnaire. Score scale 0-100 with 100 indicating a higher reported quality of life across seven different categories (seizure worry, overall quality of life, social functioning, emotional wellbeing, medication effects, energy/fatigue, and cognitive functioning).
Time Frame: 2 Years
Population: as for outcome 2
Measure: Median (Full Range); unit: QOLIE Score (0-100)
Arm/Group | NeuroBlate LITT Treatment
Number analyzed (Participants) | 2
QOLIE Score (0-100)
  Baseline QOLIE | 53.91 [26.14 to 81.68]
  24 Month QOLIE | 57.88 [34.7 to 81.06]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of patient consent (prior to the surgical procedure) to study withdraw/completion, up to 24 months.
Description: A planned study sample size of thirty (30) enrolled and treated subjects would allow events that have a 5% probability per-subject an approximately 80% chance of being observed in at least one subject in the study. Due to the inability to enroll in the FLARE study and early termination, there are insufficient data regarding adverse event rates. The two (2) reported events are captured for the patients who underwent LITT.
Arm/Group | NeuroBlate LITT Treatment
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NeuroBlate LITT Treatment (N=2)
Tinnitus (Nervous system disorders) | 1 (1)
Infection (Gastrointestinal disorders) | 1 (1) — Appendix removal

LIMITATIONS AND CAVEATS:
The per-protocol analysis was not completed because the study was terminated early and data was insufficient for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT02820740/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT02820740/SAP_002.pdf